CLINICAL TRIAL: NCT05126602
Title: Vitamin D Supplementation and Changes of Hematology Parameter, Coagulation Profile, and Clinical Improvement Among COVID-19 Patients
Brief Title: Vitamin D Supplementation and Clinical Improvement in COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bumi Herman (Other)
Responsible Party: Sponsor-Investigator, Bumi Herman, Assistant Lecturer, Hasanuddin University
Organization: Hasanuddin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0411212204
Record Dates: First submitted 2021-11-12; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: COVID-19
Keywords: Vitamin D; Hematology parameter; COVID-19; PCR Conversion; D-Dimer; Clinical Recovery
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: Two arms trial will be conducted with one group receiving a high dose of vitamin D3 whereas comparison group receiving a low dose of vitamin D3
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Masking for participants is conducted by preparing a similar chewing tablet (appearance including the color and taste). The care provider will not aware as the tablet has been unpacked. Outcome assessors are unaware of the allocation and only statistician knows the allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Dose Vitamin D3 (Experimental): A chewing tablet of 5000 IU of vitamin D3 is given twice daily, orally in the morning and evening for two weeks
  Interventions: Dietary Supplement: Vitamin D3 10000 IU
- Low Dose Vitamin D3 (Active Comparator): A chewing tablet of 1000 IU of vitamin D3 is given once daily, orally in the morning for two weeks
  Interventions: Dietary Supplement: Vitamin D3 1000 IU

INTERVENTIONS:
Dietary Supplement: Vitamin D3 10000 IU — Tablet of 5000 IU of vitamin D3 given twice daily
  Other Names: Hi-D Cholecalciferol 5000
  Arms: High Dose Vitamin D3
Dietary Supplement: Vitamin D3 1000 IU — Tablet of 1000 IU of vitamin D3 given once daily
  Other Names: Hi-D Cholecalciferol 1000
  Arms: Low Dose Vitamin D3

SUMMARY:
Background and objective Vitamin D is important as the interaction between vitamin D and its receptors at the immune cells stimulates innate and adaptive immunity. Deficiency in vitamin D is associated with increased susceptibility to infection and it is commonly found in Indonesia. Several studies indicate the potential of vitamin D supplementation against Coronavirus Disease 2019 (COVID-19), particularly in combating the proinflammatory situation as well as coagulopathy. This study aims to evaluate the supplementation of vitamin D in COVID 19 patients, particularly the changes in hematology parameters and other clinical parameters.

Method A double-blind randomized clinical trial is conducted among moderate COVID 19 patients. High-dose of vitamin D is given orally in the intervention group, compared with a low dose of vitamin D. Hematology parameters, D Dimer, conversion time on Polymerase Chain Reaction (PCR) test, and clinical symptoms are assessed

Hypothesis High Dose vitamin D shows a better hematology parameter, short PCR conversion time, and faster clinical recovery

DETAILED DESCRIPTION:
Population:

The COVID 19 patients admitted to hospital with moderate severity, defined as Individuals who show evidence of lower respiratory disease during clinical assessment or imaging and who have an oxygen saturation (SpO2) ≥94% on room air at sea level.

Methodology:

A double-blind randomized clinical trial allocated with simple random sampling

Intervention:

5000 International unit/ IU of vitamin D3 (Cholecalciferol) given orally twice daily (total 10000 IU per day)

Comparison group:

1000 International unit/ IU of vitamin D3 (Cholecalciferol) given once daily

Variables to be collected :

* The level of 25-hydroxyvitamin D in the blood
* D-Dimer
* Platelet-to-Lymphocyte Ratio (PLR)
* Total Lymphocyte Count (TLC)
* Neutrophil to Lymphocyte Ratio (NLR)
* Age
* Sex
* Comorbidities including chronic diseases
* Body Mass Index
* Handgrips Strength
* Anticoagulant administration
* Clinical Symptoms and days to recover
* Length of Stay
* Time to PCR conversion where the PCR is conducted every two days

Sample size and recruitment

Following the study in Saudi Arabia, the sample size was derived from the days to achieve recovery, where the group who received the 5000 D had an average recovery day of 6.2 ± 0.8. The intervention is expected to shorten the average recovery days up to 10%. Using the difference between the two means, the effect size derived from this result is 0.775. With 5% type 1 error and 90% power and equal allocation (1:1), the number needed for each group is 30 participants

Participants are allocated consecutively according to the permutation of the simple random sampling.

Proposed statistical analysis

1. Descriptive statistics
2. Repeated measures ANOVA
3. a Linear mixed model or generalized estimated equation will be applied to adjust the variables in the baseline

ELIGIBILITY:
1. Inclusion Criteria:

   1. Belongs to moderate case
   2. Diagnosed using PCR test
   3. Showing a vitamin D deficiency (<30 ng/dL).
2. Exclusion Criteria

   1. Pregnant or doing breastfeeding
   2. Patient under specific medication (Tuberculosis, or HIV, or malignancy) or undergo hemodialysis
   3. Receive vitamin D supplementation prior to allocation.
   4. Tested negative less than 5 days after receiving vitamin D
   5. Creatinine >2,0 mg/dL
   6. Blood Calcium >10,5 mg/dL.
   7. Ventilated
   8. Hypersensitive to vitamin D
   9. Consistent desaturation <85% with oxygen supplementation and require High-Flow Nasal Cannula (HFNC)/Extracorporeal membrane Oxygenation (ECMO) via a ventilator.
   10. Refuse to attend blood examination for follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Clinical Recovery Time | from baseline to the time when the symptoms disappear, assessed for up to 3 months
  Defined as the time where the clinical symptoms resolve completely (including cough and other symptoms of pneumonia)
Length of Stay | from the admission time to the time of hospital discharge, assessed for up to 3 months
  Defined as the duration of receiving hospital care
PCR Conversion time | from the time of diagnosis until proven negative in PCR test, assessed for up to 3 months
  Defined as the duration of the time to obtain negative result on PCR
Platelet to Lymphocyte Ratio / PLR in blood | Changes of PLR value from baseline to one week
  Defined as the ratio of platelet divided by lymphocyte value. A value of >180 indicates worse prognosis
Total Lymphocyte Count (TLC) in blood | Changes of TLC value from baseline to one week
  Defined as the ratio of platelet divided by lymphocyte value. A value of less 2000 cell/ mm3 defined as depletion and indicates worse prognosis
Neutrophil-Lymphocyte Ratio (NLR) in blood | Changes of TLC value from baseline to one week
  Defined as the ratio of Neutrophil divided by lymphocyte value. A value of less than 3.13 indicates worse prognosis
D-Dimer | Changes of D-dimer value from baseline to one week
  The D-dimer indicates the degree of fibrin degradation that is associated with blood clot breakage. A value of >500 ug/L indicates worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sisca Agustia, MD, Principal Investigator — Hasanuddin University; Amirah Faisal, MD, Principal Investigator — Hasanuddin University; Zahratul Fajri, Principal Investigator — Hasanuddin University; Nurpudji Taslim, Prof, Principal Investigator — Hasanuddin University; Suryani Armyn, Prof, Principal Investigator — Hasanuddin University; Haerani Rasyid, Prof, Principal Investigator — Hasanuddin University; Agussalim Bukhari, Prof, Principal Investigator — Hasanuddin University; Irawaty Djaharuddin, Prof, Principal Investigator — Hasanuddin University
Locations (1):
- Wahidin Sudirohusodo General Hospital, Makassar, South Sulawesi, Indonesia

IPD SHARING:
Plan to Share IPD: No
No data sharing will be done

REFERENCES:
- [Background] Ali N. Role of vitamin D in preventing of COVID-19 infection, progression and severity. J Infect Public Health. 2020 Oct;13(10):1373-1380. doi: 10.1016/j.jiph.2020.06.021. Epub 2020 Jun 20. PMID 32605780
- [Background] Meltzer DO, Best TJ, Zhang H, Vokes T, Arora V, Solway J. Association of Vitamin D Status and Other Clinical Characteristics With COVID-19 Test Results. JAMA Netw Open. 2020 Sep 1;3(9):e2019722. doi: 10.1001/jamanetworkopen.2020.19722. PMID 32880651
- [Background] Yang AP, Liu JP, Tao WQ, Li HM. The diagnostic and predictive role of NLR, d-NLR and PLR in COVID-19 patients. Int Immunopharmacol. 2020 Jul;84:106504. doi: 10.1016/j.intimp.2020.106504. Epub 2020 Apr 13. PMID 32304994
- [Background] Yao Y, Cao J, Wang Q, Shi Q, Liu K, Luo Z, Chen X, Chen S, Yu K, Huang Z, Hu B. D-dimer as a biomarker for disease severity and mortality in COVID-19 patients: a case control study. J Intensive Care. 2020 Jul 10;8:49. doi: 10.1186/s40560-020-00466-z. eCollection 2020. PMID 32665858